CLINICAL TRIAL: NCT01477242
Title: The Effect of Oral Ondansetron During Intramuscular Ketamine Use in Children
Brief Title: The Effect of Ondansetron During Intramuscular Ketamine Use in Children: A Trial in Emergency Department
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Asan Medical Center (Other); Myongji Hospital (Other)
Responsible Party: Principal Investigator, Do Kyun Kim, assistant professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-1105-114-364
Record Dates: First submitted 2011-10-23; First posted 2011-11-22 (Estimated); Last update posted 2012-01-20 (Estimated); Status verified 2012-01

CONDITIONS: Sedation and Analgesia; Side Effect of Drug
Keywords: vomiting; anti-emetics; ketamine; sedation
MeSH Terms: conditions — Agnosia; Vomiting | interventions — Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ondansetron (Experimental): Ondansetron use group
  Interventions: Drug: Ondansetron
- Placebo (Placebo Comparator): Placebo group
  Interventions: Drug: Ondansetron

INTERVENTIONS:
Drug: Ondansetron — 2mg (5mL) in < 15 kg and 4mg (10mL) in 15kg to 30kg
  Other Names: Zofran zydis; vomiset

SUMMARY:
The purpose of this study is to evaluate the anti-emetic effect of oral ondansetron. For this evaluation, the investigators will perform a multi-center, double-blind, placebo-controled, randomized study. The investigators assumption is that oral ondansetron prior to intramuscular ketamine will reduce the occurrence of ketamine-induced vomiting.

DETAILED DESCRIPTION:
Methods

* a multi-center, double-blind, placebo-controled, randomized study ( 4 tertiary hospital ED)
* survey for the occurrence of vomiting at ED and after discharge

Primary outcome

* the number of vomiting at ED and at home

Secondary outcome

* parent's satisfaction and ED length of stay

ELIGIBILITY:
Inclusion Criteria:

* children under 18 years of age
* children who are planned to admit ketamine intramuscular injection
* children with ASA classification class I or II

Exclusion Criteria:

* don't want to enroll to study
* children with condition of contraindication of ketamine (IICP, IIOP, psychosis, brain tumor, thyroid disease, porphyria)
* children with condition of contraindication of ondansetron (hypersensitivity to 5-HT3 antagonist, Long QT syndrome, severe liver failure, obstructive ileus)
* children under 3 months of age
* children whose weight are over 30 kg
* children managed by other drug with ketamine

Min Age: 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 266 (Estimated)
Dates: Start 2011-11; Primary Completion 2012-05 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
vomiting at ED stay and 12 hours after discharge | the participants will be followed for the duration of ED stay (upto 24hr) and 12hours after discharge

SECONDARY OUTCOMES:
parent's satisfaction | satisfaction will be surveyed within 48hours after discharge
length of emergency department stay | length of stay will be calculated upto 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Do Kyun Kim, M.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea